CLINICAL TRIAL: NCT03927209
Title: A Phase I, Open-label, Positron Emission Tomography Study in Healthy Male Subjects to Explore the Inhibition of Monoamine Oxidase B in the Brain After Multiple Oral Doses of BI 1467335 (Non-randomized, Open-label, Parallel-group Study)
Brief Title: A Study in Healthy Men to Test the Effects of Different Doses of BI 1467335 on MAO-B Activity in the Brain.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1386-0022; 2018-003745-41 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1467335 (low dose) (Experimental)
  Interventions: Drug: BI 1467335
- BI 1467335 (high dose) (Experimental)
  Interventions: Drug: BI 1467335

INTERVENTIONS:
Drug: BI 1467335 — tablet

SUMMARY:
The main objective of this trial is to investigate the effect of multiple oral dosing of high dose BI 1467335 over 28 days and multiple oral dosing of low dose BI 1467335 over 42 days on MAO-B occupancy in the brain compared to baseline using [11C]-L-deprenyl-D2 PET tracer in healthy male subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 21 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Non-smoker with no history of smoking
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication. Adequate methods are:

  * Condoms plus use of hormonal contraception by the female partner that started at least 2 months prior to administration of trial medication (e.g., implants, injectables, combined oral or vaginal contraceptives, intrauterine device) or
  * Condoms plus surgical sterilization (vasectomy at least 1 year prior to enrolment) or
  * Condoms plus surgically sterilised partner (including hysterectomy) or
  * Condoms plus intrauterine device or
  * Condoms plus partner of non-childbearing potential (including homosexual men) Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 90 days or within 5 half-lives, whichever is longer, of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Alcohol abuse (consumption of more than 30 g per day for males) within the 24 months prior to dosing
* Drug abuse within the 24 months prior to dosing or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Structural brain abnormality has been shown on an Magnetic Resonance Imaging (MRI)
* Severe anxiety of enclosed spaces
* Contraindication for arterial cannulation: Allen's test indicating potential risk in placement of the arterial cannula.
* Contraindication to MRI as determined by screening and safety questionnaire including but not limited to significant tattoos (as determined by the radiographer), cardiac pacemakers, aneurysm clips and cochlear implants.
* Unable to lie flat on the MRI or Positron emission tomography (PET) scanner for a prolonged period of time.
* Prior participation in other research protocols in the past year such that the total effective dose including this study would exceed 10 mSv.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwick Park Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase I trial was conducted using a non-randomised, non-controlled, open-label, parallel-group, multiple-dose design.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 1467335 10 Milligram (mg): Oral administration of 10 milligram (mg) BI 1467335 (2 film-coated tablet of 5 mg) per day for 28 days together with 240 milliliter (mL) of water.
- BI 1467335 3 Milligram (mg): Oral administration of 3 milligram (mg) BI 1467335 (3 film-coated tablet of 1 mg) per day for 42 days together with 240 milliliter (mL) of water.
Period: Overall Study
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (7.7) | 39.0 (11.4) | 41.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Reduction in Whole Brain Monoamine Oxidase (MAO)-B Availability Assessed by Positron Emission Tomography (PET) Imaging
Description: The primary endpoint of the trial was the percent reduction in whole brain MAO-B availability, as assessed by PET imaging, on the last day of treatment with BI 1467335 (Day 28 for the 10 mg dose group and Day 42 for the 3 mg dose group) compared with baseline. Image analysis was used to generate the outcome parameter for the PET data (proportional to the target availability at each PET scan) using the PET emission and the metabolite corrected arterial plasma input function in an appropriate kinetic model.
Time Frame: Baseline (day -14 to -2) and last day of treatment (Day 28 for the 10 mg dose group and Day 42 for the 3 mg dose group).
Population: PET set (PETS): This set included all subjects who were randomized and treated with at least one dose of study drug for whom at least 1 PET scan at baseline and 1 on-treatment scan were provided.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg)
Number analyzed (Participants) | 5 | 4
Percent reduction | 72.58 (11.81) | 2.43 (6.05)

2. Secondary Outcome: Percent Reduction in MAO-B Availability on Day 14 of Treatment With 10 mg BI 1467335 Compared With Baseline
Description: Percent reduction in MAO-B availability on Day 14 of treatment with 10 mg BI 1467335 compared with baseline. Image analysis was used to generate the outcome parameter for the PET data (proportional to the target availability at each PET scan) using the PET emission and the metabolite corrected arterial plasma input function in an appropriate kinetic model.
Time Frame: Baseline (day -14 to -2) and Day 14 of treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | BI 1467335 10 Milligram (mg)
Number analyzed (Participants) | 5
Percent reduction | 44.56 (16.20)

3. Secondary Outcome: Reduction in MAO-B Availability on Day 28 of Treatment With 3 mg BI 1467335 Compared With Baseline
Description: Reduction in MAO-B availability on Day 28 of treatment with 3 mg BI 1467335 compared with baseline. Image analysis was used to generate the outcome parameter for the PET data (proportional to the target availability at each PET scan) using the PET emission and the metabolite corrected arterial plasma input function in an appropriate kinetic model.
Time Frame: Baseline (day -14 to -2) and Day 28 of treatment.
Population: PET set (PETS): This set included all subjects who were randomized and treated with at least one dose of study drug for whom at least 1 PET scan at baseline and 1 on-treatment scan were provided. One subject in the 3 mg dose group was excluded from the PET analysis because had no measurement of MAO-B availability on Day 28.
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | BI 1467335 3 Milligram (mg)
Number analyzed (Participants) | 3
Percent reduction | -1.43 (6.29)

4. Secondary Outcome: MAO-B Inhibition in Platelet Rich Plasma Compared With Baseline
Description: MAO-B activity in plasma was assessed after 14 days of dosing with BI 1467335 (10 mg dose group only), 28 days of dosing (10 and 3 mg dose groups), and 42 days of dosing (3 mg dose group only).
Time Frame: Baseline (day -14 to -2) and last day of treatment (Day 28 for the 10 mg dose group and Day 42 for the 3 mg dose group).
Population: Due to missing baseline values, processing errors and errors in the conduct of the analytical assay most subjects were excluded. The small amount of available data precluded accurate evaluation of the pharmacokinetic - pharmacodynamic (PK-PD) relationship.
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Maximum Measured Concentration of BI 1467335 in Plasma
Description: Maximum measured concentration of BI 1467335 in Plasma (Cmax).
Time Frame: Within 3 hours (h) before and 20 minutes (min), 45 min, 1h, 1h 30 min, 3h, 4h, 7h, 11h, 24h (~30 min before next scheduled dosing where applicable) after administration of BI 1467335.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects in the TS for whom at least 1 PK endpoint was provided, and who were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol per liter
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg)
Number analyzed (Participants) | 5 | 5
nanomol per liter
  Day 14: number analyzed (Participants) | 5 | 0
  Day 14 | 36.4 (65.2) |
  Day 28 | 48.4 (85.3) | 2.28 (76.0)
  Day 42: number analyzed (Participants) | 0 | 5
  Day 42 |  | 3.60 (146)

6. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Time 24 h (AUC 0-24)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time 24 h.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol * hours per liter
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg)
Number analyzed (Participants) | 5 | 5
nanomol * hours per liter
  Day 14: number analyzed (Participants) | 5 | 0
  Day 14 | 85.7 (75.5) |
  Day 28: number analyzed (Participants) | 5 | 4
  Day 28 | 235 (148.0) | 4.65 (54.9)
  Day 42: number analyzed (Participants) | 0 | 5
  Day 42 |  | 4.34 (132)

ADVERSE EVENTS:
Time Frame: From the date/time of first administration of BI 1467335 until 12 a.m. on the day after subjects end of participation date. (Up to 36 days for 10mg group, up to 50 days for 3mg group)
Description: Treated set (TS): The TS included all subjects who were randomized and treated with at least one dose of study drug.
Groups:
- Total on Treatment: Total of the over all on-treatment phases of BI 1467335.
Arm/Group | BI 1467335 10 Milligram (mg) | BI 1467335 3 Milligram (mg) | Total on Treatment
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 5/5 | 3/5 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1467335 10 Milligram (mg) (N=5) | BI 1467335 3 Milligram (mg) (N=5) | Total on Treatment (N=10)
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Catheter site bruise (General disorders) | 1 | 1 | 2
Catheter site erythema (General disorders) | 0 | 1 | 1
Catheter site pain (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Feeling hot (General disorders) | 1 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT03927209/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03927209/SAP_001.pdf